CLINICAL TRIAL: NCT00560937
Title: Pilot Study of Pregnenolone Augmentation Targeting Cognitive Symptoms in Persistently Symptomatic Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Christine E. Marx, MD, Durham Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VA IRB# 00924
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2010-12-28 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Pregnenolone; Cognition; Negative Symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Pregnenolone
  Interventions: Drug: Pregnenolone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone 50 mg twice a day (BID) x 2 weeks, Pregnenolone 150 mg BID x 2 weeks, Pregnenolone 250 mg BID x 4 weeks
  Arms: 1
Drug: Placebo — Placebo (similar to active comparator) 50 mg BID x 2 weeks, Placebo (similar to active comparator) 150 mg BID x 2 weeks, Placebo (similar to active comparator) 250 mg BID x 4 weeks
  Arms: 2

SUMMARY:
This is a pilot study of pregnenolone as an augmentation treatment for schizophrenia. The goal of this placebo-controlled study is to provide preliminary efficacy data for potential pregnenolone effects on cognitive symptoms and negative symptoms in patients with schizophrenia. Depressive symptoms and positive symptoms will also be assessed.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age, any ethnic group, either sex
2. Diagnostic and Statistical Manual, 4th edition (DSM IV) diagnosis of schizophrenia or schizoaffective disorder
3. Ability to participate fully in the informed consent process, or have a legal guardian able to participate in the informed consent process.
4. Patient cohort enriched for moderate to severe cognitive symptoms (composite Brief Assessment of Cognition in Schizophrenia (BACS) score 0-3 SD below the mean).
5. No change in antipsychotic for 8 weeks or longer. No change in antipsychotic dose for 4 weeks or longer.
6. No change in anticholinergic, benzodiazepine, or mood stabilizer medications for 4 weeks or longer.
7. No anticipated need to alter any of the above medications (antipsychotics, anticholinergics, benzodiazepines, or mood stabilizers) for the 10-week duration of the study.

Exclusion Criteria:

1. Unstable medical illness or neurologic illness (seizures, cerebrovascular accident); history of prostate, breast, uterine, or ovarian cancer.
2. Use of oral contraceptives or other hormonal supplementation such as estrogen.
3. Other concomitant medications for medical conditions will be addressed on a case-by-case base to determine if exclusionary.
4. Active expression of suicidal or homicidal ideation.
5. Comorbid substance dependence (other than nicotine dependence), or presenting symptoms likely substance-induced, as judged by a study physician.
6. Female patients who are pregnant or breast-feeding.
7. Known allergy to study medication.
8. Drugs with a narrow therapeutic index (e.g. thioridazine, mesoridazine, ziprasidone, clozapine, etc) will be excluded as suggested by the Federal Drug Administration (FDA); patients taking these agents will not be eligible for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD, MA, Principal Investigator — Durham VAMC
Locations (1):
- Durham VAMC, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred between 8-05 and 4-06 for this single-site study at the Durham VAMC, Durham, NC.
Pre-assignment Details: Following the screening visit, patients were withdrawn during the placebo lead-in phase and were not randomized for the following reasons: 1. hyponatremia, 2. hospitalization, 3.pneumonia, 4.no show for follow-up study visit, 5.chest pain, 6. elevated prolactin at baseline, 7.prolonged QTc at baseline
Groups:
- Pregnenolone: * Pregnenolone 100 mg in divided doses (50 mg BID) for 2 weeks, then
  * Pregnenolone 300 mg in divided doses (150 mg BID) for 2 weeks, then
  * Pregnenolone 500 mg in divided doses (250 mg BID) for 4 weeks.
- Placebo: Placebo dosing and tablets were identical to Pregnenolone.
Period: Overall Study
Arm/Group | Pregnenolone | Placebo
Started | 10 | 11
Completed | 9 (One participant was withdrawn after 6 weeks and data were carried forward) | 9
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 10 | 11 | 21.0
  >=65 years | 0 | 0 | 0.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6) | 49 (12) | 51 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2.0
  Male | 9 | 10 | 19.0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21.0

OUTCOME MEASURES:

1. Primary Outcome: Mean Score on the Scale for the Assessment of Negative Symptoms (SANS), p=0.048
Description: The SANS assesses negative symptoms in schizophrenia. The SANS consists of 21 clinical interview questions assessing negative symptoms of schizophrenia. Each question is rated on a scale of 0 (no symptoms) to 7 (severe symptoms).
Time Frame: SANS scores at baseline and 8 weeks post-randomization (at least 4 weeks; last observation carried forward)
Population: Pilot proof of concept study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale | -10.38 (10.18) | -2.33 (4.42)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; T-test of change scores, pregnenolone vs. placebo post-treatment compared to baseline; Test type: Superiority or Other; p = .048, t-test, 2 sided

2. Secondary Outcome: Mean Score Change in Calgary Depression Scale for Schizophrenia (CDSS)
Description: The CDSS is used measure to investigate depressive symptoms in schizophrenia. The measure includes 9 questions ranked from 0 (no symptoms) to 3 (severe symptoms). Range of possible scores: 0-27.
Time Frame: Change in CDSS scores at baseline and 8 weeks (at least 4 weeks; last observation carried forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | -1.57 (2.15) | -2.00 (3.66)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.79, t-test, 2 sided

3. Primary Outcome: Mean Change of Z-scores on the Brief Assessment of Cognition in Schizophrenia (BACS)
Description: The BACS includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3.
Time Frame: Change in composite BACS scores at baseline and 8 weeks post-randomization (at least 4 weeks; last observation carried forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 0.60 (0.78) | 0.22 (0.47)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

4. Primary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS)
Description: The MATRICS is a battery for the assessment of cognitive symptoms in patients with schizophrenia. Composite T-scores are calculated (T-score ranges are -20 to +80, and are normed on gender and age). Higher scores are indicative of better cognitive performance, lower scores are indicative of poorer cognitive performance.
Time Frame: Change in composite MATRICS scores at baseline and 8 weeks post-randomization (at least 4 weeks; last observation carried forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 7.00 (8.87) | 7.00 (4.95)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; T-test of change scores, pregnenolone compared to placebo post-treatment vs. pre-randomization; Test type: Superiority or Other; p = 1.0, t-test, 2 sided

5. Secondary Outcome: Clinical Global Impression Scale (CGI-I)
Description: The CGI-I is a commonly used psychiatric scale to assess overall general improvement. The CGI-I consists of one interviewer-rated question on a scale of 1-7. Lower scores are indicative of fewer symptoms; while higher scores are indicative of more symptoms.
Time Frame: CGI-I scores at 8 weeks post-randomization (at least 4 weeks; last observation carried forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | 2.11 (0.33) | 2.89 (0.78)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.014, t-test, 2 sided

6. Secondary Outcome: Mean Score on the Positive and Negative Symptom Scale (PANSS)
Description: The PANSS is a widely used measure with several subdomains, including positive symptoms, negative symptoms, and general psychopathology of schizophrenia. Lower scores are indicative of fewer symptoms; higher scores are indicative of more symptoms. Total PANSS scores range from 0-20.
Time Frame: Change in PANSS scores at baseline and 8 weeks post-randomization (at least 4 weeks; last observation carried forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | -9.88 (9.23) | -5.44 (5.27)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during each study visit (study visits occurred every two weeks, a total of 5 study visits) for the duration of the 10 week study (following a 2 week placebo lead-in).
Description: Hillside Adverse Event Questionnaire used to obtain Adverse Events.
Arm/Group | Pregnenolone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnenolone (N=9) | Placebo (N=9)
Disorientation (date, address, mayor, MD name) (Psychiatric disorders) | 2 (3) | 2 (2)
Decreased interest in sex (General disorders) | 1 (3) | 2 (3)
Hypertension (Cardiac disorders) | 1 (2) | 1 (3)
Impaired sexual performance (General disorders) | 0 (0) | 1 (3)
Excitation/agitation (General disorders) | 0 (0) | 1 (4)
Dry Mouth (General disorders) | 1 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Restlessness (General disorders) | 2 (5) | 0 (0)
Muscle pain/stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cold extremities (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes